CLINICAL TRIAL: NCT04556136
Title: A Pilot Feasibility Study Comparing a Novel Phototherapy Kiosk to Supplementation to Promote Vitamin D Sufficiency
Brief Title: Comparing a Novel Phototherapy Kiosk to Oral Vitamin D Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Madigan Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Mary S McCarthy, Senior Nurse Scientist, Madigan Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 217121
Record Dates: First submitted 2020-07-10; First posted 2020-09-21 (Actual); Results first posted 2024-03-12 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Hypovitaminosis D
Keywords: VitaminD; UVBPhototherapy; Military
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Vitamin D

STUDY DESIGN:
Intervention Model Description: For volunteers assigned to the phototherapy kiosk, a measured dose of UVB was administered under conditions of full body exposure of 0.6 minimal erythemal dose (MED) every other week for 10 weeks. The stimulation of cutaneous vitamin D and subsequent 25(OH)D production from phototherapy was compared to the effect of a Recommended Daily Allowance (RDA) based dose of 600 IU vitamin D3 supplement daily for 10 weeks.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: A computer-generated block design was created by an onsite biostatistician and used by the research pharmacist to randomize subjects. Once a subject met the inclusion criteria, the pharmacist was notified and she relayed the group assignment to the Project Coordinator. The study team had no knowledge of the group assignment in advance.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Standing Phototherapy Kiosk (SPK) (Experimental): Volunteers assigned to this group were administered phototherapy treatments in a standing phototherapy kiosk once every other week, for 10 weeks. The treatment usually lasts no more than 10 minutes and is based on the Fitzpatrick skin type classification tool, which is self-reported via the computer touch screen in the kiosk.
  Interventions: Device: Standing Phototherapy Kiosk
- Oral Supplement (Active Comparator): Volunteers assigned to this group were provided with a 10-week supply (70 pills) of a vitamin D3 supplement. Consented subjects were instructed to take one 600 IU pill by mouth each day for ten weeks. They were instructed to take this with a meal. This dose is the RDA for adults between 18 and 70 years old according to the Institute of Medicine Committee to Review Dietary Reference Intakes for Vitamin D and Calcium.
  Interventions: Dietary Supplement: D3 Oral supplement

INTERVENTIONS:
Device: Standing Phototherapy Kiosk — Benesol is a freestanding booth designed to deliver a small amount of targeted UVB with an interactive user interface and cloud-based software that enables patient self-care. The treatment delivery mechanism uses a metal halide lamp with a series of filters and a lens to optimize full-body exposure to the narrow spectrum (293 - 303nm) of UVB light most efficient at producing vitamin D3. The device uses software to identify patients, establish individual skin types and determine dosage. The system has been designed to manage exposure time and frequency and deliver 60% of a skin-type-adjusted Minimal Erythemal Dose (MED). The expected result for users is a rise in blood levels of 25(OH)D via the endogenous pathway.
  Other Names: Phototherapy Booth
  Arms: Standing Phototherapy Kiosk (SPK)
Dietary Supplement: D3 Oral supplement — Each subject assigned to the comparison group was instructed to take one vitamin D3 pill, dispensed by the research pharmacist, each day with a meal for 70 days. Subjects were instructed not to take any additional vitamin D supplementation during the study period. This dosing frequency is consistent with the RDA recommendation. Subjects were instructed to bring their pill bottle with them when returning for their follow up appointment.
  Other Names: Vitamin D
  Arms: Oral Supplement

SUMMARY:
The purpose of this project is to demonstrate the capability of a standing phototherapy kiosk (SPK) to stimulate cutaneous vitamin D3 and subsequent production of 25 Hydroxyvitamin (OH) D safely and as efficiently as an oral vitamin D3 supplement of 600 IU taken daily over a 10 week intervention period. We will conduct a randomized controlled trial with two treatment arms; ~120 volunteers will be assigned to either the SPK or to a 600 IU daily oral vitamin D3 supplement for 10 weeks. The SPK is an innovative, networked, self-care technology that stimulates endogenous vitamin D production with two ~2-minute treatments per month. It will be tested in an ambulatory setting where enrolled/assigned participants of various baseline levels of 25(OH)D will present for a treatment dose, based on Fitzpatrick skin type category, every other week for 10 weeks. The SPK does not produce a cosmetic tan or dispense pills.

DETAILED DESCRIPTION:
The proposed pilot study uses a prospective, longitudinal, randomized design with repeated measures to address vitamin D sufficiency in Active Duty (AD), retiree, beneficiary, and Department of Army civilian populations. It is important and necessary to conduct this study with adult humans, military personnel in particular, to determine acceptability and feasibility of this phototherapy kiosk as an addition to existing Warfighter resources to promote health and resilience. Anticipating 20% attrition, approximately 120 volunteers will be recruited from Madigan Army Medical Center and Joint Base Lewis-McChord (JBLM), a large joint base in the Pacific Northwest, where over 25,000 Soldiers and Airmen train every day and regional beneficiaries number ~98,000. Recruiting efforts will attempt to capture a representative sample of the population including genders, diverse ethnicities, and a range of age (18-70 years) and body mass index, who have no contraindication for Ultraviolet (UV) B exposure or oral vitamin D supplementation. Using a computer-generated block design, volunteers will be randomized to one of two treatment groups; 1) oral vitamin D supplementation, or 2) standing phototherapy kiosk (SPK) with UVB exposure, for a 10 week period.

Group 1- Supplement: A Madigan Army Medical Center (MAMC) Research Pharmacist will dispense a 10-week supply of the vitamin D3 600 International Units (IU) oral supplement to subjects assigned to this group one time. The Project Coordinator will work with the pharmacist to coordinate pick-up of supplement bottles for subjects or optimal in-person dispensing times.

Group 2 - SPK: The Project Coordinator will oversee the phototherapy treatment. Spectrum isolation modules in the kiosk will deliver the UVB dose under supervised conditions over a 2-5 minute interval based on the Fitzpatrick skin type category with the subject wearing minimal or no clothing, preferably no more than a bathing suit and protective eye-wear. The experience in the SPK is designed to be comfortable.

We will enroll all eligible adult volunteers regardless of their baseline 25(OH)D level; it is important to show there is no potential for harm from phototherapy, even if the baseline 25(OH)D level is above 30 ng/mL. We also must learn the trajectory of vitamin D absorption and availability over a 3-4 month period in order to make evidence-based therapeutic recommendations. It is not possible to blind the subjects or research team to the group assignment. Serum levels of 25(OH)D, calcium, and parathyroid hormone will be drawn at baseline (T0), and immediately following the intervention at 10 weeks (T6); at 14 weeks (T8), 25(OH) D will be drawn to document sustainment of treatment effect. A survey will be completed at T1 to capture relevant demographic, medical history, sun exposure, travel, daily activities, and dietary data. Active duty participants will also report the number of days on profile for the previous three months, at T1 and T6. A survey regarding Device Usability will be administered upon kiosk protocol completion. We will analyze data using repeated measures analysis of variance adjusting for significant covariates such as 25(OH)D level at baseline. Logistic regression analyses will be used to predict outcomes and explain the interrelationships among variables, i.e. age, gender, body fat, BMI, ethnicity, and sun exposure relationship to 25(OH)D serum levels.

Outcomes:

1. Serum 25(OH)D level. This primary outcome will be crucial to establishing whether the device, a standing phototherapy kiosk (SPK), is equivalent to oral vitamin D3 supplementation which is currently the standard of care prescribed by licensed providers to address vitamin D insufficiency/deficiency. We will establish a baseline 25(OH)D level for both study arms.
2. Change in serum 25(OH)D at 10 weeks to reflect adequacy of SPK and supplement treatment.
3. Change in serum 25(OH)D at 14 weeks will evaluate sustainment of the post-SPK treatment level.
4. Device acceptability by Device Usability Scale. To properly evaluate the outcome of acceptability of this demonstration project involving two arms, one an SPK and the other an oral vitamin D supplement, the research team will administer the Device Usability Scale upon study completion at 14 weeks.
5. Device feasibility will be assessed by meticulously tracking of the number of potential participants screened, the number of enrolled subjects, and attrition from each arm. Reasons for attrition will be documented following a discussion with the subject, if possible.

ELIGIBILITY:
Inclusion Criteria:

* Adults, age 18 - 69 years
* Ability to read and understand English
* Subjectively in good health
* Able to stand without assistance for ~10 minutes

Exclusion Criteria:

* Any volunteer with relocation, deployment, or release from active duty in the next 4 months
* Pregnant, or currently breastfeeding, females
* Anyone with chronic health problems (e.g. kidney disease, liver disease, intestinal malabsorption)
* Any volunteer currently taking vitamin D supplementation
* Taking medications for an endocrine disorder, such as Synthroid or oral hypoglycemic agents
* Sarcoidosis
* Medications having a high potential for interaction with vitamin D:

anti-seizure medications, cyclosporine, indinavir (Crixivan) • Adults diagnosed with light allergies: Actinic prurigo, Polymorphous light eruption, Solar urticaria

• Adults diagnosed with light sensitivities: Protoporphyria, Photodermatitis, Xeroderma pigmentosum, Lupus erythematosus, Actinic dermatitis, UV-sensitive syndrome

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2018-04-30 (Actual); Primary Completion 2019-01-22 (Actual); Study Completion 2019-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary S McCarthy, PhD, Principal Investigator — Nurse Scientist, CNSCI
Locations (1):
- Madigan Army Medical Center, Tacoma, Washington, United States

REFERENCES:
- [Background] Koutkia P, Lu Z, Chen TC, Holick MF. Treatment of vitamin D deficiency due to Crohn's disease with tanning bed ultraviolet B radiation. Gastroenterology. 2001 Dec;121(6):1485-8. doi: 10.1053/gast.2001.29686. PMID 11729127
- [Background] He CS, Aw Yong XH, Walsh NP, Gleeson M. Is there an optimal vitamin D status for immunity in athletes and military personnel? Exerc Immunol Rev. 2016;22:42-64. PMID 26853300
- [Background] Holick MF, Binkley NC, Bischoff-Ferrari HA, Gordon CM, Hanley DA, Heaney RP, Murad MH, Weaver CM; Endocrine Society. Evaluation, treatment, and prevention of vitamin D deficiency: an Endocrine Society clinical practice guideline. J Clin Endocrinol Metab. 2011 Jul;96(7):1911-30. doi: 10.1210/jc.2011-0385. Epub 2011 Jun 6. PMID 21646368
- [Background] Chen TC, Chimeh F, Lu Z, Mathieu J, Person KS, Zhang A, Kohn N, Martinello S, Berkowitz R, Holick MF. Factors that influence the cutaneous synthesis and dietary sources of vitamin D. Arch Biochem Biophys. 2007 Apr 15;460(2):213-7. doi: 10.1016/j.abb.2006.12.017. Epub 2007 Jan 8. PMID 17254541
- [Background] Fitzpatrick TB. The validity and practicality of sun-reactive skin types I through VI. Arch Dermatol. 1988 Jun;124(6):869-71. doi: 10.1001/archderm.124.6.869. No abstract available. PMID 3377516
- [Background] Bogh MK, Schmedes AV, Philipsen PA, Thieden E, Wulf HC. A small suberythemal ultraviolet B dose every second week is sufficient to maintain summer vitamin D levels: a randomized controlled trial. Br J Dermatol. 2012 Feb;166(2):430-3. doi: 10.1111/j.1365-2133.2011.10697.x. PMID 22013924

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruiting efforts attempted to capture a representative sample of the population including both genders, diverse ethnicities, and a range of age (18-70 years) and BMI, who have no contraindication for UVB exposure or oral vitamin D supplementation. In addition to walk-in volunteers who read medical center flyers or social media posts, or were informed through word-of-mouth, the team attended the military base Newcomer's Orientation monthly. Recruitment period 8 months.
Pre-assignment Details: No pre-assignment activities.
Period: Overall Study
Arm/Group | Standing Phototherapy Kiosk (SPK) | Oral Supplement
Started | 53 | 53
Completed | 43 | 45
Not Completed | 10 | 8
Not completed — Lost to Follow-up | 6 | 6
Not completed — Physician Decision | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standing Phototherapy Kiosk (SPK) | Oral Supplement | Total
Number analyzed (Participants) | 53 | 53 | 106
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 52 | 49 | 101
  >=65 years | 1 | 4 | 5
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Attrition resulted in the loss of 10 participants from the Kiosk Group and 8 participants from the Oral Supplement Group.
  Participants
    number analyzed (Participants) | 43 | 45 | 88
    Female | 32 | 25 | 57
    Male | 11 | 20 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Attrition resulted in the loss of 8 participants from the Oral Supplement Grp and 10 participants from the Kiosk Grp.
  Participants
    number analyzed (Participants) | 43 | 45 | 88
    Hispanic or Latino | 7 | 8 | 15
    Not Hispanic or Latino | 36 | 37 | 73
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Due to attrition, the number analyzed is different from the number enrolled.
  Participants
    number analyzed (Participants) | 43 | 45 | 88
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 5 | 7 | 12
    White | 27 | 20 | 47
    More than one race | 7 | 8 | 15
    Unknown or Not Reported | 4 | 10 | 14
Region of Enrollment [Number; unit: participants] — Population: Due to attrition, the number analyzed differs from the number enrolled.
  participants
    United States: number analyzed (Participants) | 43 | 45 | 88
    United States | 43 | 45 | 88
Marital status [Count of Participants; unit: Participants] — Marital status obtained via demographic questionnaire; subject was asked whether he/she was single or married. Population: Due to attrition, the number of subjects analyzed differs from the number enrolled.
  Participants
    number analyzed (Participants) | 43 | 45 | 88
    Single | 8 | 12 | 20
    Married | 35 | 33 | 68
Military affiliation [Count of Participants; unit: Participants] — Subjects answered the question of military affiliation as active duty, retired or former service member, family member, none. Population: Due to attrition, the number of subjects analyzed differs from the number enrolle.
  Participants
    number analyzed (Participants) | 43 | 45 | 88
    Active duty | 22 | 28 | 50
    Retired or prior service | 11 | 8 | 19
    Family member | 8 | 6 | 14
    None | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Serum Vitamin D Level
Description: 25 Hydroxyvitamin D level in the blood
Time Frame: 10 weeks
Population: Final sample included 43 in SPK and 45 in Oral Supplement group; 10 subjects of 98 enrolled dropped out prior to the end of the study.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Standing Phototherapy Kiosk (SPK) | Oral Supplement
Number analyzed (Participants) | 43 | 45
ng/mL | 30.0 [25.8 to 37.0] | 25.5 [21.0 to 29.8]
Statistical Analysis 1: Comparison: Standing Phototherapy Kiosk (SPK) vs Oral Supplement; The intent-to-treat analysis plan was carried out with all available subject data points. No interim analysis was performed. Exploratory data analyses were conducted on serum vitamin D levels of participants assigned to either the oral supplementation or kiosk group. Analysis was restricted to participants with valid baseline serum vitamin D data and at least one follow-up blood draw. The Shapiro-Wilk test was used to assess the normality of the data distribution; Test type: Non-Inferiority — This non-inferiority study was designed to demonstrate the ability of the phototherapy kiosk to safely administer UVB radiation to participants with varying levels of 25(OH)D and achieve comparable levels of serum 25(OH)D in a similar population of adults randomized to receive RDA of 600 IU vitamin D oral supplementation daily. It is important to evaluate device equivalence to standard of care in the maintenance of sufficient levels of vitamin D in adults 18 - 70 years old; p = 0.01, Wilcoxon (Mann-Whitney) — Threshold for significance <0.05; Effect sizes for significant differences were included as eta squared (ŋ2) values

2. Primary Outcome: Change in Serum Vitamin D Level From Baseline to Week 14
Description: Change over time in 25(OH)D from baseline to week 14 in kiosk group versus supplement group.
Time Frame: Baseline and 14 weeks
Population: Final sample included 43 in SPK group and 45 in Oral supplement group; 10 of 98 dropped out
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Standing Phototherapy Kiosk (SPK) | Oral Supplement
Number analyzed (Participants) | 43 | 45
ng/mL | 27 [22.0 to 32.5] | 21 [17.0 to 30.0]

3. Primary Outcome: Percentage of Participants With Adherence
Description: Percentage of participants with adherence to daily supplement, and Percentage of phototherapy treatments received.
  Adherence to daily supplement was calculated as the percentage of participants who consumed all 70 pills.
  Adherence to phototherapy treatments was calculated as the percentage of participants who received all 6 treatments according to protocol.
Time Frame: 10 weeks
Population: Intent-to-treat analysis used to assess number consuming all of the Oral supplement and the number receiving all 6 phototherapy (SPK) treatments.
Measure: Number; unit: percentage of participants
Arm/Group | Standing Phototherapy Kiosk (SPK) | Oral Supplement
Number analyzed (Participants) | 43 | 45
percentage of participants | 98 | 98

4. Secondary Outcome: Device Acceptability Using Device Usability Scale
Description: User acceptability and satisfaction with the novel kiosk on the Device Usability Scale (DUS), also referred to as System Usability Scale. The DUS was administered to the SPK Group upon completion of the study to assess user acceptability of the intervention. This 12-item Likert-type scale assessed cleanliness, ease of use, and comfort of the kiosk with a Likert-type scale where 1= Strongly disagree to 5 = Strongly agree. Minimum score = 12, maximum score = 60. Higher scores indicate greater acceptability and satisfaction with the device.
Time Frame: 14 weeks
Population: Only the SPK group was asked about acceptability and satisfaction with the kiosk.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standing Phototherapy Kiosk (SPK) | Oral Supplement
Number analyzed (Participants) | 43 | 0
score on a scale | 55.38 (4.33) |

5. Secondary Outcome: Number of Subjects Retained at 14 Weeks
Description: We examined the number of subjects remaining at 14 weeks.
Time Frame: Baseline to 14 weeks
Population: Subject retention at the 14-week measurement point
Measure: Count of Participants; unit: Participants
Arm/Group | Standing Phototherapy Kiosk (SPK) | Oral Supplement
Number analyzed (Participants) | 39 | 41
Participants | 39 | 41

ADVERSE EVENTS:
Time Frame: The study was 11 months in length.
Description: Participants in the Phototherapy group were asked to report skin reactions (eg sunburn) due to exposure from the phototherapy kiosk. Erythema events that resembled an E3 or E4 as characterized in "Chapter 5 of Radiation dosimetry: physical and biological aspects" were defined as adverse events. In the Supplement group, taking more of the D3 supplement than prescribed could be harmful.
Arm/Group | Standing Phototherapy Kiosk (SPK) | Oral Supplement
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/53
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/53
Other Adverse Events (participants affected / at risk) | 0/53 | 0/53

LIMITATIONS AND CAVEATS:
Due to the use of an untested device, the appropriate sample size was estimated based on previous and current vitamin D studies, involving an adult population, and a similar approach to vitamin D supplementation. Study conducted at a single center in a geographic location known for limited opportunity for exposure to UVB as a source for vitamin D therefore low vitamin D status is common. Results may not be generalizable to adults in communities throughout the US.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-27): https://cdn.clinicaltrials.gov/large-docs/36/NCT04556136/Prot_SAP_001.pdf